CLINICAL TRIAL: NCT01898676
Title: An Open Label, Randomized, Four-period, Two-sequence, Fully Replicated, Single-dose, Crossover Study of the Relative Bioavailability of Two Formulations of Extended-release Divalproex Sodium Tablets in Fed Patients With Stable Epilepsy.
Brief Title: A Study in Stable Epilepsy Patients Comparing Brand and Generic Divalproex Sodium Extended Release Tablets
Acronym: Epilepsy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vince & Associates Clinical Research, Inc. (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RIHSC #13-019D
Record Dates: First submitted 2013-06-17; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-06

CONDITIONS: Epilepsy
Keywords: Extended-release divalproex sodium; Depakote ER
MeSH Terms: conditions — Epilepsy | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Divalproex Sodium Extended Release 250mg (Active Comparator): Treatment A: A single 2-tablet dose of divalproex sodium extended-release tablet, 250mg. Each subject will have 2 treatments with this medication and two treatments with a single 2-tablet dose of DEPAKOTE 250mg tablet.
  Interventions: Drug: Divalproex Sodium Extended-release 250mg; Drug: DEPAKOTE 250mg
- DEPAKOTE 250mg (Active Comparator): Treatment B: A single 2-tablet dose of DEPAKOTE ER tablet, 250mg. Each subject will have 2 treament period with this medication and 2 treatment periods with a single 2-tablet dose of Divalproex Sodium Extended-Release 250mg tablet.
  Interventions: Drug: Divalproex Sodium Extended-release 250mg; Drug: DEPAKOTE 250mg

INTERVENTIONS:
Drug: Divalproex Sodium Extended-release 250mg — Two tablets of Divalproex Sodium Extended-Release 250mg will be given to the subject in two treatment periods
  Other Names: DEPAKOTE 250mg
Drug: DEPAKOTE 250mg — Two tablets of DEPAKOTE 250mg will be given to the subject in two treatment periods.
  Other Names: Divalproex Sodium Extended-Release 250mg

SUMMARY:
A study in stable epilepsy patients comparing levels of valproic acid after administration of brand and generic divalproex sodium extended release tablets.

DETAILED DESCRIPTION:
Study consists of a screening visit, four treatment periods and a final follow-up visit. Each treatment period consists of a four night in-house stay followed by two outpatient visits. Each treatment period will be separated by a washout period. During each treatment period, safety evaluations will include vital signs, physical exams, safety laboratory tests, weight measurement, electrocardiograms, adverse event collection and concomitant medication recording. Pharmacokinetic blood samples will be collected during each treatment period. Seizure activity will be recorded in a seizure diary during the study. A standardized high-fat, high-calorie meal will be served prior to each dose during each treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand, sign and date the informed consent form
* Male or female 18 to 55 years old with a diagnosis of epilepsy who are stable
* Body mass 18 to 34 kg/m, inclusive
* Is continuously receiving a fixed dose of their AED medication(s)for a minimum of 30 days prior to screening
* Stay on the same dosages of their routine concomitant medications throughout the study
* Healthy, as determined by pre-study medical history, vital signs, physical exam, ECG and the opinion of the investigator
* Normal renal function per laboratory test
* No clinically relevant labs.
* Negative for hepatitis B, C and HIV
* For females, negative pregnancy test
* Negative for drugs of abuse and alcohol
* Nonsmoker or has not smoked within the past six months.
* Some over-the-counter medications may be permitted at the discretion of the investigator
* Able to communicate well and comply with study procedures, requirements and restrictions

Exclusion Criteria:

* History or presence of clinically significant medical disorders
* Have a current psychiatric disorder
* History of status epilepticus within 90 days of screening
* Any other condition that the investigator would feel could interfere with the safety of the subject or the study protocol.
* Taking three or more AED medications
* Use of felbamate, aspirin, carbapenem antibiotics, rifampin, ritonavir, macrolide antibiotics, cholestyramine, and/or risperidone.
* Use of any investigational agent or medical device within 30 days of screening.
* History of clinically significant drug allergy that in the opinion of the investigator may compromise the subject's safety or study results.
* History of known hypersensitivity to divalproex sodium or its excipients
* History of alcohol or drug abuse or dependence in the past 5 years
* Consumed alcohol, caffeine or other xanthine-containing foods or beverages within 48 hours prior to each clinic admission.
* Consumed grapefruit and/or grapefruit containing products within days prior to admission to the clinic on Day -1 and they agree not to consume grapefruit and/or grapefruit containing products for the duration of their study involvement
* Participated in any strenuous physical exercise within 72 hours before admission to the clinic on Day 1 and agrees to abstain from the duration of their study involvement.
* Acute illness at screening and/or at admission to the clinic
* Lactose intolerance or unusual dietary habits.
* Blood donation within 8 weeks of admission to this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate generic divalproex sodium extended release to Depakote ER | Approximately 2.5 months
  This is an open-label, randomized, two-sequence, two-treatment, single dose, four-period, fully replicated crossover study in which 16 subjects will receive one of the two study drugs, Depakote ER or a generic equivalent, during each treatment period. Subjects will be patients with epilepsy who are otherwise healthy and who are stable on anti-epileptic therapy, not including any formulation of divalproex sodium.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley D. Vince, DO, Principal Investigator — Vince & Associates Clinical Research, Inc.
Locations (1):
- Vince & Associates Clinical Research, Inc., Overland Park, Kansas, United States